CLINICAL TRIAL: NCT02557867
Title: The Effect of Obesity in Dexmedetomidine Metabolic Clearance
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 14-253; 1150197 (Other Grant/Funding Number: FONDECYT)
Record Dates: First submitted 2015-09-06; First posted 2015-09-23 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Obesity
Keywords: dexmedetomidine; pharmacokinetic; obesity
MeSH Terms: conditions — Obesity | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obese (Experimental): Body composition measurement before surgery using Dual energy X-ray absorptiometry. Dexmedetomidine infusion during surgery. Venous blood sampling for dexmedetomidine plasmatic levels during and after surgery. Liver blood flow indirect non-invasive assessment after surgery using indocyanine. Liver biopsy during surgery.
  Interventions: Drug: Dexmedetomidine
- Non-obese (Experimental): Body composition measurement before surgery using Dual energy X-ray absorptiometry. Dexmedetomidine infusion during surgery. Venous blood sampling for dexmedetomidine plasmatic levels during and after surgery. Liver blood flow indirect non-invasive assessment after surgery using indocyanine. Liver biopsy during surgery.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 0.5 μg/kg over 10 minutes and then, 0.5 mcg/kg/h throughout surgery.
  Other Names: Precedex

SUMMARY:
The purpose of this study is to study the effect of obesity in dexmedetomidine pharmacokinetics and pharmacodynamic profile.

DETAILED DESCRIPTION:
The investigators expect to find an inverse correlation between the amount of fat mass and liver blood flow or with the enzymatic metabolic capacity. Results will be based on a population pharmacokinetic modeling analysis performed in NONMEM program. The investigators will first account for the effect of different measured size scalars on volumes and clearances and then they will search for plausible covariates (liver blood flow, enzymatic capacity, degree of hepatic steatosis, etc) on dexmedetomidine metabolic clearance. A pharmacokinetic model capable of characterizing clearance changes in the obese using more plausible biological covariates will be tried to be defined.

ELIGIBILITY:
Inclusion Criteria for obese patients:

* American Society of Anesthesiology classification I-III patients.
* Both genders.
* Age between 18 - 60 years.
* Body mass index higher than 40 Kg/m2.

Inclusion Criteria for non-obese patients:

* American Society of Anesthesiology classification I-II patients
* Both genders.
* Age between 18 - 60 years
* Body mass index lower than 30 Kg/m2.

Exclusion Criteria:

* Known allergy to study drugs
* Uncontrolled hypertension.
* Heart block greater than first degree.
* Chronic hepatic and kidney disease.
* Patients taking any drug acting in the central nervous system within 24 hrs before surgery.
* Patients taking drugs that induce overexpression of liver cytochrome P450-complex enzymes (Carbamazepine, Phenytoin, Phenobarbital, Rifampicin, Dexamethasone, Griseofulvin, Terbinafine, Prednisone, Hydrocortisone, Modafinil).)
* Known addiction to illicit drugs.
* Pregnancy.
* Current or past oncologic disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Dexmedetomidine plasmatic levels | From start of infusion (min): 5, 10, 20, 30, 45, 60, 90, 120, 150, 180; from end of infusion (min): 5, 10, 20, 30, 60, 90, 120, 240, 360, 720
  Measured by high performance liquid chromatography

SECONDARY OUTCOMES:
Steatohepatitis score | 3 months after liver biopsy specimen collection
  Using liver biopsy, a score for steatohepatitis will be applied on samples from all patients
Plasma disappearance rate of indocyanine | 2 hours after arrival to Post-Anesthesia Care Unit
  Using indocyanine green and LiMON monitor (Pulsion Medical Systems) surrogate measures of liver blood flow will be registered.
Enzyme expression | 3 months after liver biopsy specimen collection
  Liver samples will be analyzed for UGT2B10 and UGT1A4 expression (involved in dexmedetomidine metabolization)
Hemodynamics | Recorded at every blood sample collection (5, 10, 20, 30, 45, 60, 90, 120, 150, 180 min) during anesthesia
  Heart rate and arterial pressure will be recorded during anesthesia
Anesthetic depth | Recorded at every blood sample collection (5, 10, 20, 30, 45, 60, 90, 120, 150, 180 min) during anesthesia
  Using a bispectral index monitor, anesthetic depth will be monitorized through out surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Luis I Cortínez, MD, Principal Investigator — Associate Professor Ordinary Category
Locations (1):
- Hospital Clinico Pontificia Universidad Catolica, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Han PY, Duffull SB, Kirkpatrick CM, Green B. Dosing in obesity: a simple solution to a big problem. Clin Pharmacol Ther. 2007 Nov;82(5):505-8. doi: 10.1038/sj.clpt.6100381. PMID 17952107
- [Background] Green B, Duffull SB. What is the best size descriptor to use for pharmacokinetic studies in the obese? Br J Clin Pharmacol. 2004 Aug;58(2):119-33. doi: 10.1111/j.1365-2125.2004.02157.x. PMID 15255794
- [Background] Casati A, Putzu M. Anesthesia in the obese patient: pharmacokinetic considerations. J Clin Anesth. 2005 Mar;17(2):134-45. doi: 10.1016/j.jclinane.2004.01.009. PMID 15809132
- [Background] Hall JE, Uhrich TD, Barney JA, Arain SR, Ebert TJ. Sedative, amnestic, and analgesic properties of small-dose dexmedetomidine infusions. Anesth Analg. 2000 Mar;90(3):699-705. doi: 10.1097/00000539-200003000-00035. PMID 10702460
- [Background] Hsu YW, Cortinez LI, Robertson KM, Keifer JC, Sum-Ping ST, Moretti EW, Young CC, Wright DR, Macleod DB, Somma J. Dexmedetomidine pharmacodynamics: part I: crossover comparison of the respiratory effects of dexmedetomidine and remifentanil in healthy volunteers. Anesthesiology. 2004 Nov;101(5):1066-76. doi: 10.1097/00000542-200411000-00005. PMID 15505441
- [Background] Gurbet A, Basagan-Mogol E, Turker G, Ugun F, Kaya FN, Ozcan B. Intraoperative infusion of dexmedetomidine reduces perioperative analgesic requirements. Can J Anaesth. 2006 Jul;53(7):646-52. doi: 10.1007/BF03021622. PMID 16803911
- [Background] Kaivosaari S, Toivonen P, Aitio O, Sipila J, Koskinen M, Salonen JS, Finel M. Regio- and stereospecific N-glucuronidation of medetomidine: the differences between UDP glucuronosyltransferase (UGT) 1A4 and UGT2B10 account for the complex kinetics of human liver microsomes. Drug Metab Dispos. 2008 Aug;36(8):1529-37. doi: 10.1124/dmd.108.021709. Epub 2008 May 12. PMID 18474681
- [Background] Bedogni G, Agosti F, De Col A, Marazzi N, Tagliaferri A, Sartorio A. Comparison of dual-energy X-ray absorptiometry, air displacement plethysmography and bioelectrical impedance analysis for the assessment of body composition in morbidly obese women. Eur J Clin Nutr. 2013 Nov;67(11):1129-32. doi: 10.1038/ejcn.2013.159. Epub 2013 Sep 11. PMID 24022260
- [Background] Brunt EM, Janney CG, Di Bisceglie AM, Neuschwander-Tetri BA, Bacon BR. Nonalcoholic steatohepatitis: a proposal for grading and staging the histological lesions. Am J Gastroenterol. 1999 Sep;94(9):2467-74. doi: 10.1111/j.1572-0241.1999.01377.x. PMID 10484010
- [Background] Li W, Zhang Z, Wu L, Tian Y, Feng S, Chen Y. Determination of dexmedetomidine in human plasma using high performance liquid chromatography coupled with tandem mass spectrometric detection: application to a pharmacokinetic study. J Pharm Biomed Anal. 2009 Dec 5;50(5):897-904. doi: 10.1016/j.jpba.2009.06.012. Epub 2009 Jun 16. PMID 19577876
- [Background] Ji QC, Zhou JY, Gonzales RJ, Gage EM, El-Shourbagy TA. Simultaneous quantitation of dexmedetomidine and glucuronide metabolites (G-Dex-1 and G-Dex-2) in human plasma utilizing liquid chromatography with tandem mass spectrometric detection. Rapid Commun Mass Spectrom. 2004;18(15):1753-60. doi: 10.1002/rcm.1548. PMID 15282775
- [Background] Duffull SB, Dooley MJ, Green B, Poole SG, Kirkpatrick CM. A standard weight descriptor for dose adjustment in the obese patient. Clin Pharmacokinet. 2004;43(15):1167-78. doi: 10.2165/00003088-200443150-00007. PMID 15568893
- [Derived] Rolle A, Paredes S, Cortinez LI, Anderson BJ, Quezada N, Solari S, Allende F, Torres J, Cabrera D, Contreras V, Carmona J, Ramirez C, Oliveros AM, Ibacache M. Dexmedetomidine metabolic clearance is not affected by fat mass in obese patients. Br J Anaesth. 2018 May;120(5):969-977. doi: 10.1016/j.bja.2018.01.040. Epub 2018 Mar 28. PMID 29661414